CLINICAL TRIAL: NCT01510782
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Doses (0.2 mg to 120 mg Administered by Intravenous Infusion and 40 mg to 120 mg Administered by Subcutaneous Injection) of BI 655064 (Buffer Solution for Injection) in Healthy Male Volunteers (Randomised, Single-blind, Placebo-controlled Within Dose Groups, Clinical Phase I Study)
Brief Title: Single Rising Dose Study (Intravenous Infusion and Subcutaneous Injection) of BI 655064 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1293.1; 2011-002251-34 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-01-12; First posted 2012-01-16 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
MeSH Terms: interventions — BI 655064

ARMS (4):
- BI 655064 subcutaneous (Experimental): Escalating single dose as solution for subcutaneous injection
  Interventions: Drug: BI 655064
- Placebo to BI 655064 subcutaneous (Placebo Comparator): Escalation single dose as solution for subcutaneous injection (Placebo)
  Interventions: Drug: Placebo to BI 655064
- BI 655064 intravenous (Experimental): Escalating single dose as solution for intravenous infusion
  Interventions: Drug: BI 655064
- Placebo to BI 655064 intravenous (Placebo Comparator): Escalating single dose as solution for intravenous infusion (Placebo)
  Interventions: Drug: Placebo to BI 655064

INTERVENTIONS:
Drug: Placebo to BI 655064 — intravenous infusion of escalating doses
  Arms: Placebo to BI 655064 intravenous
Drug: Placebo to BI 655064 — subcutaneous injection of escalating doses
  Arms: Placebo to BI 655064 subcutaneous
Drug: BI 655064 — intravenous infusion of escalating doses
  Arms: BI 655064 intravenous
Drug: BI 655064 — subcutaneous injection of escalating doses
  Arms: BI 655064 subcutaneous

SUMMARY:
To investigate safety and tolerability of BI 655064 in healthy male volunteers following intravenous infusion of escalating single doses and following subcutaneous injection. Exploration of the pharmacokinetics and pharmacodynamics of BI 655064 after single dosing and determination of the bioavailability of subcutaneous injections of BI 655064.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Changes in vital signs (blood pressure [BP], pulse rate [PR]) | up to 70 days post treatment
Changes in 12-lead ECG (electrocardiogram) | up to 70 days post treatment
Incidence of adverse events | up to 70 days post treatment
Assessment of global tolerability by investigator | up to 70 days post treatment
Assessment of local tolerability by investigator | up to 70 days post treatment

SECONDARY OUTCOMES:
Maximum measured concentration of the analyte in plasma | up to 1656 hours post treatment
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity | up to 1656 hours post treatment
Area under the concentration-time curve of the analyte in the plasma over the time interval from 0 to the last measurable time point of the dose | up to 1656 hours post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1293.1.1 Boehringer Ingelheim Investigational Site, Berlin, Germany

REFERENCES:
- [Derived] Albach FN, Wagner F, Huser A, Igel J, Joseph D, Hilbert J, Schoelch C, Padula SJ, Steffgen J. Safety, pharmacokinetics and pharmacodynamics of single rising doses of BI 655064, an antagonistic anti-CD40 antibody in healthy subjects: a potential novel treatment for autoimmune diseases. Eur J Clin Pharmacol. 2018 Feb;74(2):161-169. doi: 10.1007/s00228-017-2362-8. Epub 2017 Nov 10. PMID 29127458